CLINICAL TRIAL: NCT06368323
Title: Effect of Community Choir Singing in People With Chronic Post-stroke Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Collaborators: Toronto Metropolitan University (Other); Université de Montréal (Other); Université du Québec à Trois-Rivières (Other); University of South Florida (Other)
Responsible Party: Principal Investigator, Anna Zumbansen, Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-01-24-9931
Record Dates: First submitted 2024-04-01; First posted 2024-04-16 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: A parallel group randomized trial design with a secondary crossover extension
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be measured by blinded assessors where possible, using blinded video or audio recordings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB Group (Experimental): First choir, then usual care
  Interventions: Behavioral: Choir singing; Other: Usual care
- BA Group (Experimental): First usual care, then choir
  Interventions: Behavioral: Choir singing; Other: Usual care

INTERVENTIONS:
Behavioral: Choir singing — The 12-week intervention will consist of 12 in-person choir-singing sessions (1 session/week, 1,5 h/session, total 18h) conducted by a choir master in addition to home training (3 x 30-minutes-sessions/week, total 18h). In total, participants will undergo the intervention for 3 hours/week for 12 weeks (i.e., 36 hours).
Other: Usual care — Rehabilitation services received by patients and social activities will be monitored and documented.

SUMMARY:
The goal of this randomized controled trial is to test the effects of assigning people with chronic post-stroke aphasia to 12 weekly choir sessions, compared to usual care.

The main question it aims to answer is:

Does the assignment to a choir singing program causes a beneficial effect on functional communication and language recovery as well as psychosocial outcomes compared to usual care in the rehabilitation of people with chronic post-stroke aphasia?

Participants will have:

12 in-person choir-singing sessions (1 session/week, 1,5 h/session, total 18h) conducted by a choir master, and home singing training (3 x 30-minutes-sessions/week, total 18h)

DETAILED DESCRIPTION:
Description of study population Additional information: Participants with chronic aphasia due to stroke will be recruited from four participating centers in Canada and the United States.

Study design Additional information: A parallel group randomized trial design with a secondary crossover extension was chosen for this study to offer the intervention to all participants. Participants will be randomized in a 1:1 ratio to two study arms (AB/BA, A = 12 weekly choir sessions and home singing training, B = usual care) stratified for aphasia severity (according to the Quick Aphasia Battery overall score), age, time since last stroke and their interest in music (according to the Barcelona Music Reward Questionnaire). Measures at the "macro" level will be collected at Baseline, Completion and 2-months Follow-up time points for each group. At the "micro" level (i.e., at choir sessions 2, 6, 10 and 12) data will be collected during as well as pre and post choir-singing.

Intervention Additional information: The repertoire in the comunity choir activity will consist of popular songs in English or French. Half of the songs will be pre-determined and half will be chosen by the choir members from a list, based on a vote during the first week of the intervention. Eligible songs will remain within the range of an octave and include a variety of tempi (but fast tempi will be slowed down if needed to facilitate word production). Depending on the group's abilities, the Choir Director will decide in which keys the songs will be performed, and whether they will be sung in unison or with simple harmonies. Songs in canon will be included in the predetermined repertoire to easily create harmonies. Each session will include (in this order): 15 minutes for vocal warm-up; 25 minutes of work on the song repertoire; 20 minutes for a social break with refreshments.

For the home training, participants will be instructed to sing at home with a video guide on an online platform. Each home training session will include (in this order): 10 minutes for vocal warm-up; and 20 minutes sing-along using songs of the repertoire. Song lyrics will be displayed on the video.

To monitor the usual care, each participant (and/or caregiver) will complete a form and/or have a weekly 5-15-minute phone/Zoom call with a research assistant to collect the usual care data including type and time spent in social activities and rehabilitation services, as well as adverse events.

Randomization and concealment For randomization, an online system will be used by a researcher not involved in data collection.

Each participant will be assigned an identification number upon inclusion in the study. After completion of the baseline assessments, the independent researcher will receive the list of participants' IDs with their stratification data (age, time post-stoke, aphasia severity, level of interest in music) to perform the randomization.

Blinding:

Outcomes will be measured by blinded assessors where possible, based on video or audio recordings.

Planned analyses:

Primary hypothesis:

Participants assigned to the choir intervention over 12 weeks will demonstrate a significantly larger improvement in macro-level measures compared to those receiving usual care.

Secondary hypothesis:

Participants who completed the choir intervention with 80% adherence over 12 weeks will demonstrate a larger improvement in macro-level measures compared to those receiving usual care.

The gains will be maintained for the participants with 80% adherence.

There will be immediate changes in micro-level measures after a choir session (Session 6).

There will be differences in pre-post-session variations of micro-level measures between Session 2, 6 and 10.

There will be differences in pre-post-session variations between the usual rehearsal (Session 10) and the Concert (Session 12).

ELIGIBILITY:
Inclusion Criteria:

* People with chronic aphasia following stroke
* English or French as language of daily use
* Last stroke must have occurred at least 6 months before the start of the first assessments in the study protocol.

Exclusion Criteria:

* Regular music making in the past 6 months
* Visual deficit that cannot be corrected and might impair testing
* Hearing deficit that cannot be corrected and might impair testing
* Presence of neurological/psychiatric co-morbidity or substance abuse
* No ability to produce vocal sound through singing/humming
* Legally considered unable to make decisions for oneself

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-04-22 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Communication Index | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  The ability to communicate one's feelings and basic needs effectively / is computed by averaging the percentage scores (score/total×100) of the Communicative Activity Log (CAL) and the communication subscale of the Stroke Impact Scale 3.0 (SIS).
  Minimum value=0; Maximum value=100; Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Level of confidence in communication | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  Individual's subjective perception of their ability to effectively communicate in various situations / assessed with the Communication Confidence Rating Scale for Aphasia (CCRSA), a self-reported assessment in 10 questions.
  Minimum value=4; Maximum value=40; Higher scores mean a better outcome.
Aphasia severity index | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  The aphasia severity index quantifies the extent of language impairment experienced by individuals with aphasia / assessed using the Quick Aphasia Battery (QAB).
  Minimum value=0; Maximum value=10; Higher scores mean a better outcome.
Speech and language in functional communication | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  The ability of an individual to effectively use verbal communication skills / assessed with a part of the AphasiaBank protocol to elicit connected speech in participants Minimum value=0; Maximum value=100; Higher scores mean a better outcome.
Apraxia of speech severity | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  The degree or level of impairment in the motor planning and execution of speech movements / assessed with the Apraxia of Speech Rating Scale (ASRS-3.5) experienced by individuals with apraxia Minimum value=0; Maximum value=52; Higher scores mean a worse outcome.
Health related quality of life assessed by the the Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  Individual's subjective perception of their physical, emotional, mental, and social well-being in relation to their health status and the impact of illness or treatment on their overall quality of life / assessed with the Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39) Minimum value=39; Maximum value=195; Higher scores mean a better outcome.
Emotional wellbeing | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  The state of an individual's mental and emotional health, encompassing their overall mood, psychological resilience, and ability to cope with stressors and life challenges / assessed using the General Health Questionnaire (GHQ-12) Minimum value=0; Maximum value=36; Higher scores mean a worse outcome.
Social participation | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  Active engagement of individuals within their community or society, involving various social activities, interactions, and roles. / assessed using the corresponding SIS participation subscale.
  Minimum value=8; Maximum value=40; Higher scores mean a better outcome.
Generic measure of health | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  Short-Form 6-Dimension version 2 (SF-6Dv2) is a survey on 6 health domains: Physical functioning, Role functioning, Pain, Vitality, Social functioning, Mental health.
  Minimum value= 0; Maximum value= 100;Higher scores mean a better outcome.
Appetence to music | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  An individual's inclination or attraction towards music / Barcelona Music Reward Questionnaire (BMRQ)
  Minimum value= 20; Maximum value= 100 ; Higher scores mean a better outcome.
Singing voice abilities | T1 (baseline, week 1), T2 (week 15), T3 (week 16), T4 (week 30), T5 (week 31)
  Overall singing voice quality, tuning and rhythmic accuracy / assessed following a standardized protocol

OTHER OUTCOMES:
Voice - Pitch | Before and afrer choir sessions 2, 6, 10 and 12
  Pitch mean, standard deviation, and range in spontaneous speech based on a quick standardized voice production protocol
Voice - Maximum Phonation Time | Before and afrer choir sessions 2, 6, 10 and 12
  Maximum Phonation Time based on a quick standardized voice production protocol
Voice - Dynamic range | Before and afrer choir sessions 2, 6, 10 and 12
  Dynamic range based on a quick standardized voice production protocol
Mood | The first and last 10 minutes of sessions 2, 6, 10 and 12 as well as the last 10 minutes of the break.
  Temporary state of mind or temper / assessed with the Observed Emotion Rating Scale (OERS), an observational tool for rating two positive emotions (pleasure and general alertness) and three negative emotions (anger, anxiety or fear, and sadness) over a defined 10-minute period. A longer display of emotion is indicated by higher scores.
Biosocial indexes | Before and afrer choir sessions 2, 6, 10 and 12
  Cortisol and oxytocin measures / measured in salivary samples
Expectations on a 100-scale | T1 (baseline, week 1),T5 (week 31)
  Measures expectations based on a feedback questionnaire. Minimum value=0; Maximum value=100; Higher scores mean a better outcome.
Satisfaction on a 100-scale | T1 (baseline, week 1),T5 (week 31)
  Measures satisfaction based on a feedback questionnaire. Minimum value=0; Maximum value=100; Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Zumbansen, PhD, Principal Investigator — University of Ottawa; Arla Good, PhD, Principal Investigator — Toronto Metropolitan University; Frank Russo, PhD, Principal Investigator — Toronto Metropolitan University; Carole Anglade, PhD, Principal Investigator — Université de Montréal; Édith Durand, PhD, Principal Investigator — Université du Québec à Trois-Rivières; Jennifer Bugos, PhD, Principal Investigator — University of South Florida
Locations (4):
- University of South Florida, Tampa, Florida, United States
- Canada (3):
  - University of Ottawa, Ottawa, Ontario
  - Toronto Metropolitan University, Toronto, Ontario
  - Université de Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siponkoski ST, Pitkaniemi A, Laitinen S, Sarkamo ER, Pentikainen E, Eloranta H, Tuomiranta L, Melkas S, Schlaug G, Sihvonen AJ, Sarkamo T. Efficacy of a multicomponent singing intervention on communication and psychosocial functioning in chronic aphasia: a randomized controlled crossover trial. Brain Commun. 2022 Dec 27;5(1):fcac337. doi: 10.1093/braincomms/fcac337. eCollection 2023. PMID 36687394
- [Background] Anna Zumbansen, Isabelle Peretz, Carole Anglade, Josée Bilodeau, Suzanne Généreux, Michelyne Hubert & Sylvie Hébert (2017) Effect of choir activity in the rehabilitation of aphasia: a blind, randomised, controlled pilot study, Aphasiology, 31:8, 879-900, DOI: 10.1080/02687038.2016.1227424
- See also: The SingWell Project — https://www.singwell.ca/

DOCUMENTS (1):
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT06368323/ICF_000.pdf